CLINICAL TRIAL: NCT00279240
Title: The Indian Diabetes Prevention Programme Shows That Lifestyle Modification and Metformin Prevent Type 2 Diabetes in Asian Indian Subjects With Impaired Glucose Tolerance (IDPP1)
Brief Title: Life Style Modifications Prevents Type 2 Diabetes in Asian Indians
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.V. Hospital for Diabetes (Other)
Allocation: Randomized | Masking: None | Purpose: Prevention
Other Study IDs: IDPP1
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Last update posted 2006-01-24 (Estimated); Status verified 2002-07

CONDITIONS: Diabetes
Keywords: Impaired glucose tolerance; Intervention; Prevention
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance | interventions — Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
Three year prospective randomised controlled trial in IGT subjects to study the effect of metformin and lifestyle modification in preventing the conversion to diabetes

DETAILED DESCRIPTION:
Lifestyle modification helps in primary prevention of diabetes in multiethnic Americans, Finnish and Chinese populations. In a prospective community based study, we tested if the conversion to diabetes could be influenced by interventions in native Asian Indians with impaired glucose tolerance (IGT) who were younger, leaner and more insulin resistant than the above populations.

We randomized 531 (Men : Women, 421 : 110) subjects with IGT [mean age of 45.9 + 5.7 years and body mass index (BMI) of 25.8 + 3.5 kg/m2 into four groups. Group 1 was the control (CON), Group 2 was advised lifestyle modification (LSM), Group 3 was treated with metformin (MET) and Group 4 with LSM plus MET. Primary outcome measure was type 2 diabetes diagnosed by the WHO criteria.

In a median follow up of 30 months, three year cumulative incidence of diabetes were 55.0%, 39.3%, 40.5% and 39.5% in group 1 to 4 respectively. The relative risk reduction was 28.5% with LSM (95 % confidence interval (CI), (20.5 - 37.3), (p=0.018), 26.4% with MET (95% CI, 19.1 - 35.1) (p = 0.029) and 28.2% with LSM plus MET (95% CI, 20.3 - 37.0), (P=0.022) versus control group. The numbers needed to treat to prevent one incident case of diabetes were 6.4 for LSM, 6.9 for MET and 6.5 for LSM+MET.

Conversion of IGT to diabetes is high in native Asian Indians. LSM and metformin significantly reduced the incidence of diabetes in Asian Indians with IGT. There was no added benefit by combining both.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female. 35 - 55 years. No Known history of diabetes. Willing and available for a three years study.

Exclusion Criteria:

* Pregnant women. Subjects with major illness such as cancer, hepatic or cardiac diseases. Tranferable jobs.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2001-03; Study Completion 2004-12

PRIMARY OUTCOMES:
Reduction in conversion of IGT to diabetes

SECONDARY OUTCOMES:
Benefits of the drug on anthropometric variables and biochemical parameters

CONTACTS AND LOCATIONS:
Overall Officials: Ambady Ramachandran, MD,PhD,DSc., Principal Investigator — Director
Locations (1):
- Diabetes Research Centre & MV Hospital for Diabetes, Chennai, Tamil Nadu, India